CLINICAL TRIAL: NCT06094192
Title: Personalized Synchronization of Cortical Rhythms to Improve Memory in Alzheimer's Disease
Brief Title: Improving Memory in Alzheimer's Disease With Noninvasive Brain Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Robert Reinhart, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 4555_2
Record Dates: First submitted 2023-10-14; First posted 2023-10-23 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active stimulation (Experimental): Memory performance data is collected during active brain stimulation and reported 1 year later
  Interventions: Device: High definition transcranial electrical current stimulation
- sham stimulation (Sham Comparator): Memory performance data is collected during sham brain stimulation and reported 1 year later
  Interventions: Device: High definition transcranial electrical current stimulation

INTERVENTIONS:
Device: High definition transcranial electrical current stimulation — Low-intensity and safe, noninvasive application of electrical current to the human scalp with the goal of gradually modulating levels of neuronal excitability.

SUMMARY:
The investigators will evaluate the theory that Alzheimer's disease-related memory impairment derives from the inefficient orchestration of rhythmic activity at the level of large-scale cortical networks. The results as expected to elucidate AD-related pathophysiology and set groundwork for the development of drug-free interventions for improving memory in AD and related dementias.

DETAILED DESCRIPTION:
The investigators hypothesize that AD-related memory impairments emerge from large-scale functional dysconnectivity, and by stimulating the brain noninvasively with extremely weak levels of electrical current, the investigators may be able to re-synchronize connectivity and stabilize or improve memory and cognitive function, measured behaviorally. The experimental intervention involves the application of low-intensity, high-definition, transcranial electrical current stimulation while subjects perform a variety of computer-based tasks that probe memory and cognitive function.

ELIGIBILITY:
All subjects. Age 50-100 years. We will equally recruit subjects with respect to gender, race, ethnicity, socioeconomic and other factors to allow the results of this research to yield the greatest generalizability.

Mild AD dementia. Meets probable AD dementia NIA-AA criteria 86; MoCA 10-25 85; performance on Uniform Data Set version 3 (UDS-3) delayed recall (Craft Story 21) and recognition (Benson Complex Figure) memory worse than 1.5 SD for age and education; worse than 1.5 SD for age and education in at least one other cognitive domain (e.g., language, executive functioning) based on other tests in the UDS-3. A summary of the NIA-AA criteria for AD dementia are that the patient has (1) dementia, such that cognitive or behavioral symptoms (a) are interfering with the ability to function at work or usual activities, (b) represent a decline from previous level of functioning, (c) are not explained by delirium or major psychiatric disorder, (d) are detected and diagnosed, and (e) involve a minimum of two domains including memory, executive function, visuospatial abilities, language, and personality or behavior or comportment; (2) insidious onset; (3) clear-cut history of worsening of cognition; (4) prominent cognitive deficits by history and examination from either (a) an amnestic presentation or (b) a non-amnestic presentation, which can be a language, visuospatial, or executive dysfunction presentation; and lastly (5) no (a) substantial concomitant cerebrovascular disease, (b) core features of Dementia with Lewy Bodies, (c) prominent features of behavioral variant frontotemporal dementia (FTD), (d) prominent features of primary progressive aphasia, or (e) evidence for another concurrent, active disorder or use of medication that could have a substantial effect on cognition. All diagnoses are made by the BU ADRC clinical core consensus and confirmed by Dr. Budson. The majority of patients will have a positive AD biomarker, either from cerebrospinal fluid (CSF) or positron emission tomography (PET). See also Additional Inclusion/Exclusion criteria below.

MCI due to AD. Meets MCI due to AD according to NIA-AA criteria 86; MoCA >18 85; performance on Uniform Data Set version 3 (UDS-3) delayed recall (Craft Story 21) and recognition (Benson Complex Figure) memory worse than 1.0 SD for age and education adjusted norms. A summary of the NIA-AA criteria for MCI due to AD are that there is (1) clinical concern reflecting a change in cognition reported by patient, informant, or clinician; (2) objective impairment in one or more domains, typically including memory; (3) preservation of independence in functional abilities; (4) not demented; (5) a rule out of vascular, traumatic, and medical causes of cognitive decline; (6) evidence of longitudinal decline in cognition, when feasible; (7) history consistent with AD genetic factors, where relevant. All diagnoses are made by the BU ADRC clinical core consensus and confirmed by Dr. Budson. The majority of patients will have a positive AD biomarker, either from CSF or PET. See also Additional Inclusion/Exclusion criteria below.

Healthy controls. Healthy controls will also be recruited from the BU ADRC and will be age, education, and gender matched to the AD patients. They will have a MoCA > 2585 and performance within 1.0 SD for age and education adjusted norms on Uniform Data Set version 3 (UDS-3). All "diagnoses" of healthy controls will be made by the BU ADRC clinical core consensus and confirmed by Dr. Budson. The majority of healthy controls will have a negative AD biomarker, either from CSF or PET. See also Additional Inclusion/Exclusion criteria below.

All subjects. Current conditions allowed: mild depression and/or anxiety not requiring hospitalization or medications other than what are listed below; hyperlipidemia; hypercholesterolemia; hypertension; heart disease; asthma; gastroesophageal reflux disease; edema; treated hypothyroidism; systemic vascular disease (but not stroke); dermatological disorders; ophthalmologic disorders. Prior conditions excluded: stroke, traumatic brain injury, other brain or systemic disorder that, in the opinion of Dr. Budson, has produced a permanent alteration of cognition. Current medications allowed: selective serotonin reuptake inhibitors; cholinesterase inhibitors (for the patients with AD); statins; beta adrenergic blockers; bronchodilators; ace inhibitors; calcium channel blockers; angiotensin II receptor blockers; other antihypertensive agents; histamine-2 receptor antagonists; proton-pump inhibitors; diuretics; thyroid medications; aspirin; non-narcotic analgesics; antiplatelet agents; vitamins & minerals; topical medications; eye drops.

Inclusion/exclusion criteria related to tasks, EEG and tACS. Subjects must have normal or corrected-to-normal vision, color vision, nonpregnant, no metal implants in head, no implanted electronic devices, no skin sensitivity, and no claustrophobia.

Additional exclusion criteria. Subjects will be excluded if they cannot understand the informed consent or the experimental procedures. Subjects will be excluded if they have a significant vision and/or hearing impairment which will prevent them from understanding the informed consent and from completing the experimental procedures.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Memory performance (active stimulation condition) | Time Frame: Memory performance data is collected during active brain stimulation and reported 1 year later
  The accuracy of task performance on memory test
Memory performance (sham stimulation condition) | Time Frame: Memory performance data is collected during sham brain stimulation and reported 1 year later
  The accuracy of task performance on memory test

CONTACTS AND LOCATIONS:
Locations (1):
- 677 Beacon St. Room 308, Boston, Massachusetts, United States